CLINICAL TRIAL: NCT01638260
Title: Liraglutide With or Without NEAT in Type 2 Diabetes Mellitus; Effects on HbA1c, Weight, Blood Pressure, Quality of Life and Health Care Costs.
Brief Title: GLP-1 and Non-exercise Activity Thermogenesis in RHZ
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated because of insufficient number of subjects included.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC 12-2-033
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: NEAT; liraglutide; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Placebo Comparator): Subjects will inject liraglutide once daily for 26 weeks
  Interventions: Drug: Liraglutide
- Liraglutide and NEAT (Active Comparator): Subjects will inject liraglutide once daily and combine this treatment with activating lifestyle, by increasing NEAT.
  Interventions: Behavioral: NEAT

INTERVENTIONS:
Drug: Liraglutide — Liraglutide once daily 1.8 mg injection subcutaneously, 26 weeks
  Arms: Liraglutide
Behavioral: NEAT — Increasing NEAT by activating lifestyle interventions, combined with liraglutide once daily 1.8mg injections subcutaneously
  Arms: Liraglutide and NEAT

SUMMARY:
- Rationale: Treatment with glucagon-like peptide 1 (GLP-1) has been shown to reduce plasma glucose levels to a further extent when added to standard therapy in type 2 diabetes mellitus. Given the well-known beneficial effects of GLP-1 analogues on glucose metabolism by stimulating insulin release, suppressing elevated glucagon levels, delaying gastric emptying and reducing food intake, it is anticipated that liraglutide developed by Novo Nordisk (Victoza®) also has beneficial effects in type 2 diabetes mellitus as has been proven by several trials. Type 2 diabetes mellitus is associated with obesity and sedentary lifestyle. Obesity occurs when energy intake exceeds energy expenditure (EE) over a period of time. It has been presumed that activity energy expenditure and daily energy expenditure are lower in most people in Western societies. Increasing non-exercise activity thermogenesis (NEAT), defined as all energy expended due to everyday activity, exclusive of volitional exercise, may be an effective way to maintain daily EE and combat overweight and obesity. One way to promote NEAT is to decrease the amount of time spent on sedentary behaviors (e.g. watching television).

This leads us to hypothesize that adding NEAT to GLP-1 analogues in type 2 diabetes has an additive effect on glucose regulation, weight control and blood pressure. On the other hand, we hypothesize that a decrease in HbA1c, weight and blood pressure could add to an improved quality of life and less health care costs. Therefore, the primary purpose of this study is to determine the synergistic effect of liraglutide and activating lifestyle by increasing NEAT on glucose metabolism and weight. First line therapy of type 2 diabetes mellitus currently consists of lifestyle changes with metformin. When failure of this regime occurs, sulfonylurea derivates and/or thiazolidinediones can be added. One third of patients with type 2 diabetes mellitus fail with this regimen after 5 years of monotherapy, and nowadays GLP-1 analogues can be added to prevent deterioration of glycaemic control. However, comparison of this strategy with NEAT has not been performed and the synergistic effect of combination of GLP-1 with increasing NEAT has not been investigated. Treatment with GLP-1 analogues in combination with NEAT could theoretically overcome all shortcomings of current treatment strategies of type 2 diabetes mellitus.

Objective:

* Primary objectives

  * To determine the change in HbA1c from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) after 26 weeks of treatment with liraglutide versus liraglutide with NEAT
  * To determine the change in weight from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) after 26 weeks of treatment with liraglutide versus liraglutide with NEAT
* Secondary objectives

  * To assess the change in blood pressure from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) after 26 weeks of treatment with liraglutide versus liraglutide with NEAT
  * To assess the change in quality of life from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) after 26 weeks of treatment with liraglutide versus liraglutide with NEAT
  * To assess the change in NEAT from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) after 26 weeks of treatment with liraglutide versus liraglutide with NEAT
  * To asses the health-care related costs at baseline, after 26 weeks of treatment with liraglutide versus liraglutide with NEAT, and after 52 weeks (end of follow-up)

Study design: Randomized controlled intervention study

- Study population: Men and women with type 2 diabetes mellitus, insufficiënt glycaemic control during maximum (tolerable) dose monotherapy with metformin or a sulfonylurea derivate or during combination therapy with metformin and a sulfonylurea derivate or a thiazolinedione, HbA1c above 7,0%, age between 40 - 75 years old, BMI above 25 kg/m2

Intervention: One group receives once daily subcutaneously liraglutide 1.8mg added to standard anti-diabetic care and the other group receives once daily subcutaneously liraglutide 1.8mg added to standard anti-diabetic care and an activating lifestyle by increasing NEAT

Main study parameters/endpoints: The main study parameter is the percent change in HbA1c and weight. Secondary study parameters are change in blood pressure, quality of life as measured using EQ-5D and SF-36 questionnaire, NEAT as measured using an activPAL™ accelerometer and cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities
* Men or women with type 2 diabetes mellitus
* Insufficiënt glycaemic control during maximum (tolerable) dose monotherapy with metformin or a sulfonylurea derivate or during combination therapy with metformin and a sulfonylurea derivate or a thiazolinedione
* HbA1c ≥ 7.0% at screening
* BMI ≥ 25.0 kg/m2 at screening
* Age between 40-75 years

Exclusion Criteria:

* Type 1 diabetes mellitus
* HbA1c ≥ 10% at screening
* Use of GLP-1 receptor agonist (exenatide, liraglutide or other) or pramlintide or any DDP-4 inhibitor within 3 months prior to screening
* Use of insulin within 3 months prior to screening
* An acute coronary or cerebrovascular event in the previous 3 months at screening
* Chronic heart failure NYHA class IV at screening
* Estimated glomerular filtration rate (eGFR) as per Modification of Diet in Renal Disease (MDRD) < 30 ml/min/1.73m2 at screening
* Liver disease, defined as alanine or aspartate aminotransferase levels more than 2.5 the upper limit of normal range at screening
* Malignant neoplasm
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or family history of medullary thyroid cancer
* Chronic or acute pancreatitis
* Abuse or dependence of alcohol or drugs (as defined by DSM-IV)
* Any acute condition or exacerbation of chronic condition that would in the investigator's opinion interfere with the study
* Known or suspected hypersensitivity or intolerance to liraglutide
* Known to be uncooperative or noncompliant
* Simultaneous participation in any other clinical study of an investigational product
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) | 6 times, screening, week 0, week 13-26-39-52
Change in weight from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) | 6 times, screening, week 0, week 13-26-39-52

SECONDARY OUTCOMES:
Change in blood pressure from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) | 6 times, screening, week 0, week 13-26-39-52
Change in quality of life from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) | 3 times, week 0, 26, 52
  Quality of life questionnaires SF-36 en EQ-5D will be used.
Change in NEAT from baseline and end of treatment (26 weeks) and end of follow-up (52 weeks) | 3 times, week 0, 26, 52
  Neat will be measured using ActivPal accelerometer during one week.
Health-care related costs | At baseline, after 26 weeks and after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas C Schaper, Prof., MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands